CLINICAL TRIAL: NCT03000257
Title: A Multicenter, Phase 1, Open-Label, Dose-Escalation Study of ABBV-181 as Monotherapy and in Combination With Another Anti-Cancer Therapy in Subjects With Advanced Solid Tumors
Brief Title: A Study of Budigalimab (ABBV-181) in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M15-891; 2016-002520-89 (EudraCT Number)
Record Dates: First submitted 2016-12-15; First posted 2016-12-22 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumors
Keywords: Budigalimab; Cancer; Advanced Solid Tumors; Non-small cell lung cancer (NSCLC); Triple negative breast cancer; Ovarian cancer; Hepatocellular carcinoma; Gastric cancer; Small cell lung cancer; Mesothelioma; Cholangiocarcinoma; Merkel cell carcinoma; Head and neck cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Hepatocellular; Stomach Neoplasms; Small Cell Lung Carcinoma; Mesothelioma; Cholangiocarcinoma; Carcinoma, Merkel Cell; Head and Neck Neoplasms | interventions — venetoclax; rovalpituzumab tesirine; budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABBV-181 plus Venetoclax (Experimental): Venetoclax will be taken once daily beginning 7 days prior to cycle 1 and continuing daily for a 28 day cycle and ABBV-181 will be administered every 4 weeks.
  Interventions: Drug: Venetoclax; Drug: ABBV-181
- ABBV-181 (Experimental): ABBV-181 will be administered at escalating dose levels in 28-day dosing cycles (2 doses per cycle). Based on available safety, pharmacokinetic, and pharmacodynamic data from the dose-escalation part of the study, participants will be enrolled in dose-expansion cohorts to further evaluate ABBV-181 at a dose level which is at or below the Maximum tolerated dose (MTD). In the Monotherapy Expansion portion of the study, ABBV-181 will be administered in 28-day dosing cycles at either 1 dose per cycle or 2 doses per cycle. Based on available safety, PK and PD data from the single agent dose-escalation part of the study, a dose for ABBV-181 will be selected to evaluate in combination with Rovalpituzumab Tesirine or venetoclax.
  Interventions: Drug: ABBV-181
- ABBV-181 plus Rovalpituzumab Tesirine (Experimental): Rovalpituzumab Tesirine will be given once every six weeks times two doses and ABBV-181 will be administered every 3 weeks.
  Interventions: Drug: Rovalpituzumab Tesirine; Drug: ABBV-181

INTERVENTIONS:
Drug: Venetoclax — Tablet taken orally
  Arms: ABBV-181 plus Venetoclax
Drug: Rovalpituzumab Tesirine — Intravenous infusion
  Arms: ABBV-181 plus Rovalpituzumab Tesirine
Drug: ABBV-181 — Intravenous infusion
  Other Names: Budigalimab

SUMMARY:
This is an open-label, Phase I, dose-escalation study to determine the recommended Phase 2 dose (RPTD), maximum tolerated dose (MTD), and evaluate the safety and pharmacokinetic (PK) profile of budigalimab. This study will also evaluate the safety and tolerability of budigalimab in combination with Rovalpituzumab Tesirine and budigalimab in combination with venetoclax. The study will consist of 3 parts: budigalimab monotherapy dose escalation and expansion, budigalimab in combination with Rovalpituzumab Tesirine and budigalimab in combination with venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have an advanced solid tumor and must not be a candidate for surgical resection or other approved therapeutic regimen known to provide clinical benefit. For dose escalation, the participant may have been previously treated with a programmed cell death 1 (PD-I) targeting agent. For dose expansion, the participant must be PD-I/PD-L1 targeting agent naïve. For Part 2 budigalimab in combination with rovalpituzumab tesirine, the participant must have SCLC with progressive disease and have failed platinum containing therapy and be PD-1/PD-L1 targeting agent naïve. For Part 3 budigalimab in combination with venetoclax, the participant must have locally advanced or metastatic NSCLC and received 1 to 4 prior lines of therapy in the advanced or metastatic setting including 1 regimen that included a PD-1 or PD-L1 targeting agent which was discontinued following disease progression. Participants who are naïve to treatment with a PD-1/PD-L1 targeting agent OR who have received more than 1 regimen containing a PD-1/PD-L1 targeting agent are NOT eligible for Part 3.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 for the monotherapy cohort and an ECOG 0 to 1 for budigalimab in combination with rovalpituzumab tesirine cohort (Part 2) and budigalimab in combination with venetoclax (Part 3).
* Participants have adequate bone marrow, renal, hepatic and coagulation function.
* Participants must have measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 in the dose escalation portion of the trial. Participants in the expansion cohort must have measurable disease per RECIST version 1.1 or disease evaluable by assessment of tumor antigens. Participants enrolled in budigalimab in combination with venetoclax cohort (Part 3) must have measurable disease per RECIST version 1.1.

Exclusion Criteria:

* Participant has received anticancer therapy including chemotherapy, immunotherapy, radiation therapy, biologic, small molecule, herbal therapy, or any investigational therapy within a period of 5 half-lives, prior to the first dose of budigalimab or Rovalpituzumab Tesirine or venetoclax.
* For budigalimab in combination with rovalpituzumab tesirine cohort (Part 2), participant must not have had prior exposure to Rovalpituzumab Tesirine or a pyrrolobenzodiazepine (PBD) based drug.
* Participant has unresolved adverse events greater than grade 1 from prior anticancer therapy except for alopecia.
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose (with certain exceptions).
* History of primary immunodeficiency, bone marrow transplantation, chronic lymphocytic leukemia, solid organ transplantation, or previous clinical diagnosis of tuberculosis.
* Confirmed positive test results for human immunodeficiency virus (HIV), or participants with chronic or active hepatitis A, B or C. Participants who have a history of hepatitis B or C who have undetectable hepatitis B (HBV) DNA or hepatitis C (HCV) RNA after anti-viral therapy may be enrolled.
* Participant has known history or inflammatory bowel disease, pneumonitis, or known uncontrolled metastases to the central nervous system (CNS) (with certain exceptions).
* Participants with a history of or ongoing pneumonitis or interstitial lung disease are also excluded.
* For budigalimab plus venetoclax therapy (Part 3), participant must not receive a strong or moderate inducer or inhibitor of cytochrome P450 (CYP)3A within 7 days before first venetoclax dose.
* For budigalimab plus venetoclax therapy (Part 3), participants with a known gastrointestinal disorder (i.e.: malabsorption syndrome), complication (i.e.: dysphagia) or surgery that could make consumption or absorption of oral medication problematic are also excluded.
* All Cohorts: Participants with a history of Stevens-Johnson syndrome (SJS), Toxic epidermal necrolysis (TEN), or drug reaction with eosinophilia and systemic symptoms (DRESS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Part 1: Recommended Phase 2 Dose (RPTD) for Budigalimab | Up to 6 months
  If a maximum tolerated dose (MTD) is reached, the RPTD of budigalimab will not be a dose higher than the defined MTD, and will be selected based on the type(s) and occurrence(s) of dose limiting toxicities which occur in addition to the MTD. If a MTD is not reached, then the RPTD will be defined based on the safety and other available data.
Part 1: Maximum tolerated dose (MTD) of Budigalimab | Up to 6 months
  MTD will be defined at the highest dose level at which less than 2 of 6 subjects or less than 33% of (if cohort is expanded beyond 6) participants experience a dose limiting toxicity.
Part 1 and Part 3: Terminal Half-life (t1/2) of Budigalimab | Up to 4 Weeks
  Terminal phase elimination half-life (t1/2) of Budigalimab
Part 1 and Part 3: Maximum Observed Serum Concentration (Cmax) of Budigalimab | Up to 12 Weeks
  Maximum Serum Concentration (Cmax) of Budigalimab
Part 1 and Part 3: Time to Cmax (Tmax) of Budigalimab | Up to 12 Weeks
  Time to maximum plasma concentration of Budigalimab
Part 1 and Part 3: Area Under the Serum Concentration Time Curve from Time 0 to Last Measurable Concentration (AUCt) of Budigalimab | Up to 12 Weeks
  Area Under the Plasma Concentration-time Curve from time 0 to last measurable concentration (AUCt) of Budigalimab
Part 2: Recommended Phase 2 Dose (RPTD) and Schedule for Budigalimab and Rovalpituzumab Tesirine Combination | Up to 6 Months
  The safety and tolerability of a single dose of Budigalimab in combination with Rovalpituzumab Tesirine will be assessed in patients with advanced small cell lung cancer (SCLC) to determine the RPTD and schedule for the combination.
Part 3: Recommended Phase 2 Dose (RPTD) and Schedule for Budigalimab and Venetoclax Combination. | Up to 6 Months
  The safety and tolerability of Budigalimab in combination with venetoclax will be assessed in patients with metastatic Non-Small Cell Lung Cancer (NSCLC) to determine the RPTD for the combination.
Part 3: Maximum Observed Serum Concentration (Cmax) for Venetoclax | Up to 12 Weeks
  Maximum Serum Concentration (Cmax) for Venetoclax
Part 3: Area Under the Serum Concentration Time Curve from Time 0 to 24 Hours Post-dose (AUC(0-24)) of Venetoclax | Up to 12 Weeks
  Area Under the Plasma Concentration-time Curve from time 0 to time 0 to 24 hours post-dose (AUC(0-24)) of Venetoclax
Part 3: Time to Cmax (Tmax) of Venetoclax | Up to 12 Weeks
  Time to maximum plasma concentration of of Venetoclax
Part 1, Part 2, Part 3: Number of Participants with Adverse Events | From first dose of study drug until 90 days following last dose of study drug (up to 24 months)
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Part 2: Terminal Half-life (t1/2) of Budigalimab | Up to 4 Weeks
  Terminal phase elimination half-life (t1/2) of Budigalimab
Part 2: Terminal Half-life (t1/2) of Rovalpituzumab Tesirine | Up to 4 Weeks
  Terminal phase elimination half-life (t1/2) of Rovalpituzumab Tesirine
Part 2: Maximum Observed Serum Concentration (Cmax) of Rovalpituzumab Tesirine | Up to 12 Weeks
  Maximum Serum Concentration (Cmax) of Rovalpituzumab Tesirine
Part 2: Area Under the Serum Concentration Time Curve from Time 0 to Last Measurable Concentration (AUCt) of Rovalpituzumab Tesirine | Up to 12 Weeks
  Area Under the Plasma Concentration-time Curve from time 0 to last measurable concentration (AUCt) of Rovalpituzumab Tesirine
Part 2: Area Under the Serum Concentration Time Curve from Time 0 to Last Measurable Concentration (AUCt) of Budigalimab | Up to 12 Weeks
  Area Under the Plasma Concentration-time Curve from time 0 to last measurable concentration (AUCt) of Budigalimab
Part 2: Time to Cmax (Tmax) of Budigalimab | Up to 12 Weeks
  Time to maximum plasma concentration of Budigalimab
Part 2: Time to Cmax (Tmax) of Rovalpituzumab Tesirine | Up to 12 Weeks
  Time to maximum plasma concentration of Rovalpituzumab Tesirine
Part 1 and Part 3: Objective response rate (ORR) | First dose of study drug through at least 30 days after last dose of study drug.
  ORR is defined as the proportion of subjects with a confirmed partial or complete response to the treatment.
Part 1 and Part 3: Clinical benefit rate (CBR, defined as CR, PR or SD) | First dose of study drug through at least 30 days after last dose of study drug.
  CBR defined as the proportion of subjects with a confirmed partial response (PR), complete response (CR), or stable disease.
Part 1 and Part 3: Progression-free survival (PFS) | First dose of study drug through at least 30 days after last dose of study drug.
  PFS time is defined as the time from the participant's first dose of study drug (Day 1) to either the participant's disease progression or death, whichever occurs first.
Part 1, Part 2 and Part 3: Duration of objective response (DOR) | First dose of study drug through at least 30 days after last dose of study drug.
  DOR for a participant is defined as the time from the participant's initial objective response to study drug therapy to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (5):
  - Moores Cancer Center at UC San Diego /ID# 157374, La Jolla, California
  - The University of Chicago Medical Center /ID# 157375, Chicago, Illinois
  - Carolina BioOncology Institute /ID# 157376, Huntersville, North Carolina
  - South Texas Accelerated Research Therapeutics /ID# 157378, San Antonio, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 157377, Fairfax, Virginia
- Australia (3):
  - Blacktown Hospital /ID# 167386, Blacktown, New South Wales
  - St Vincent's Hospital Melbourne /ID# 167552, Fitzroy Melbourne, Victoria
  - Linear Clinical Research /ID# 170797, Nedlands, Western Australia
- Medizinische Universitaet Graz /ID# 168752, Graz, Styria, Austria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen /ID# 170702, Edegem, Antwerpen
  - UZ Gent /ID# 170881, Ghent, Oost-Vlaanderen
- Cross Cancer Institute /ID# 167603, Edmonton, Alberta, Canada
- Finland (2):
  - Tampere University Hospital /ID# 166839, Tampere, Pirkanmaa
  - Docrates Cancer Center /ID# 166838, Helsinki
- France (4):
  - Institut Bergonie /ID# 162662, Bordeaux, Gironde
  - Institut du Cancer de Montpellier - Val d'Aurelle /ID# 163999, Montpellier, Herault
  - Centre Leon Berard /ID# 162660, Lyon, Rhone
  - Institut Gustave Roussy /ID# 162753, Villejuif, Val-de-Marne
- Japan (3):
  - National Cancer Center Hospital East /ID# 166433, Kashiwa-shi, Chiba
  - National Hospital Organization Kyushu Cancer Center /ID# 206229, Fukuoka, Fukuoka
  - National Cancer Center Hospital /ID# 166279, Chuo-ku, Tokyo
- Spain (3):
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 163862, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 163861, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 163925, Valencia
- Taiwan (2):
  - National Taiwan University Hospital /ID# 163997, Taipei
  - Taipei Medical University Hospital /ID# 163998, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambert SL, Zhang C, Guo C, Turan T, Masica DL, Englert S, Fang Y, Sheridan J, McLaughlin RT, Tribouley C, Vosganian G, Afar D. Association of Baseline and Pharmacodynamic Biomarkers With Outcomes in Patients Treated With the PD-1 Inhibitor Budigalimab. J Immunother. 2022 Apr 1;45(3):167-179. doi: 10.1097/CJI.0000000000000408. PMID 35034046
- [Derived] Calvo E, Spira A, Miguel M, Kondo S, Gazzah A, Millward M, Prenen H, Rottey S, Warburton L, Alanko T, Cassier PA, Yoh K, Italiano A, Moreno V, Peltola K, Seto T, Toyozawa R, Afar DE, Englert S, Komarnitsky P, Lambert S, Parikh A, Vosganian G, Gao B. Safety, pharmacokinetics, and efficacy of budigalimab with rovalpituzumab tesirine in patients with small cell lung cancer. Cancer Treat Res Commun. 2021;28:100405. doi: 10.1016/j.ctarc.2021.100405. Epub 2021 May 25. PMID 34329846
- [Derived] Italiano A, Cassier PA, Lin CC, Alanko T, Peltola KJ, Gazzah A, Shiah HS, Calvo E, Cervantes A, Roda D, Tosi D, Gao B, Millward M, Warburton L, Tanner M, Englert S, Lambert S, Parikh A, Afar DE, Vosganian G, Moreno V. First-in-human phase 1 study of budigalimab, an anti-PD-1 inhibitor, in patients with non-small cell lung cancer and head and neck squamous cell carcinoma. Cancer Immunol Immunother. 2022 Feb;71(2):417-431. doi: 10.1007/s00262-021-02973-w. Epub 2021 Jul 3. PMID 34216247
- [Derived] Powderly J, Spira A, Kondo S, Doi T, Luke JJ, Rasco D, Gao B, Tanner M, Cassier PA, Gazzah A, Italiano A, Tosi D, Afar DE, Parikh A, Engelhardt B, Englert S, Lambert SL, Kasichayanula S, Mensing S, Menon R, Vosganian G, Tolcher A. Model Informed Dosing Regimen and Phase I Results of the Anti-PD-1 Antibody Budigalimab (ABBV-181). Clin Transl Sci. 2021 Jan;14(1):277-287. doi: 10.1111/cts.12855. Epub 2020 Dec 26. PMID 32770720